CLINICAL TRIAL: NCT06533930
Title: Evaluation of the Relationship Between Optic Nerve Diameter and Optic Nerve Sheath Diameter Measured by Transorbital Sonography With Clinical, Radiological, and Electrophysiological Parameters in Multiple Sclerosis Patients
Status: Completed | Type: Observational
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Mustafa Çetiner, Associate Professor, Kutahya Health Sciences University
Other Study IDs: 2023/11-27
Record Dates: First submitted 2024-07-30; First posted 2024-08-01 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Transorbital Sonography; Optic Nerve Sheath Diameter; Optic Nerve Diameter; Magnetic Resonance Imaging; Visual Evoked Potentials; Optical Coherence Tomography
MeSH Terms: conditions — Multiple Sclerosis | interventions — Evoked Potentials, Visual; Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients with Multiple Sclerosis: (MS Patients)
  Interventions: Other: Transorbital Sonography; Other: Orbita Magnetic Resonance Imaging; Other: Visual Evoked Potentials; Other: Optical Coherence Tomography
- Healthy Controls (HC): Healthy Controls (HC)
  Interventions: Other: Transorbital Sonography

INTERVENTIONS:
Other: Transorbital Sonography — OND and ONSD of participants in the MS patient group and healthy control group were measured by TOS.
  Other Names: TOS
Other: Orbita Magnetic Resonance Imaging — OND and ONSD of participants in the MS patient group were measured by orbita MRI.
  Other Names: MRI
  Groups: Patients with Multiple Sclerosis
Other: Visual Evoked Potentials — P100 amplitude and P100 latency values of participants in the MS patient group were measured by VEP.
  Other Names: VEP
  Groups: Patients with Multiple Sclerosis
Other: Optical Coherence Tomography — pRNFL thickness of participants in the MS patient group were measured by OCT.
  Other Names: OCT
  Groups: Patients with Multiple Sclerosis

SUMMARY:
The primary aim of this study is to evaluate the reliability of optic nerve diameter (OND) and optic nerve sheath diameter (ONSD) measurements made with transorbital sonography (TOS) and magnetic resonance imaging (MRI) in patient groups that may progress with subclinical optic atrophy over time, such as those with multiple sclerosis (MS). The secondary aims of this study are to compare the relationship of TOS with visual evoked potentials (VEP) and optical coherence tomography (OCT) parameters used in the assessment of the afferent visual pathway in MS and its clinical subtypes and to evaluate the potential of TOS as a diagnostic and monitoring tool for detecting optic nerve atrophy, subclinical axonal loss, and clinical disability in MS.

DETAILED DESCRIPTION:
The study included 102 patients with MS-81 with relapsing-remitting MS (RRMS), 19 with secondary progressive MS (SPMS), and 2 with primary progressive MS (PPMS)-as well as 34 healthy controls, all selected according to the inclusion and exclusion criteria. Demographic data for all participants, and clinical characteristics of the MS patient group, were recorded. Expanded Disability Status Scale (EDSS) measurements were performed for the patients. Then, TOS, orbital MRI, VEP and OCT examinations were applied to the individuals in the patient group on the same day for each eye. Measurements recorded included OND and ONSD by TOS and MRI, P100 latency and amplitude by VEP, and peripapillary retinal nerve fiber layer (pRNFL) thickness by OCT. In the healthy control group, OND and ONSD were measured using only transorbital TOS to establish normal measurement ranges.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-65
* Having been diagnosed with Multiple Sclerosis
* Undergoing disease-modifying therapy (DMT) for more than 6 months
* EDSS score ≤ 7

Exclusion Criteria:

* Patients whose Multiple Sclerosis diagnosis is uncertain
* Having ocular pathology that may affect optic nerve measurements (e.g., glaucoma, high myopia, history of ocular surgery)
* Having major systemic diseases that may affect optic nerve measurements (e.g., diabetes mellitus, hypertension)
* EDSS score > 7
* Having experienced a clinical relapse or optic neuritis within the last 6 months.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients having been diagnosed with MS and healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Transorbital Sonography | 2 minutes
  OND and ONSD of participants in the MS patient group and healthy control group were measured by TOS.
Orbita Magnetic Resonance Imaging | 30 minutes
  OND and ONSD of participants in the MS patient group were measured by orbita MRI.

SECONDARY OUTCOMES:
Visual Evoked Potentials | 20 minutes
  Visual Evoked Potentials
Optical Coherence Tomography | 15 minutes
  pRNFL thickness of participants in the MS patient group were measured by OCT.
Expanded Disability Status Scale | 30 minutes
  Disability Status Evaluation. A score of 0 on the scale indicates normal neurological status, while a score of 10 means MS-related death.

CONTACTS AND LOCATIONS:
Locations (1):
- Kutahya Health Sciences University, Faculty of Medicine, Kütahya, Kütahya, Turkey (Türkiye)